CLINICAL TRIAL: NCT01496001
Title: The Effect of Tumor - Breast Volume Ratio on Cosmetic and Functional Outcomes in Breast Conserving Surgery Patients; a Prospective Cohort Study
Brief Title: Cosmetic and Functional Outcomes After Breast Conserving Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Dr. Zoltan Matrai, Principal Investigator, National Institute of Oncology, Hungary
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NIO-BCS-QoL
Record Dates: First submitted 2011-12-12; First posted 2011-12-21 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Early unilateral breast cancer
MeSH Terms: conditions — Breast Neoplasms; Unilateral Breast Neoplasms | interventions — Mastectomy, Segmental; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cohort (Experimental)
  Interventions: Procedure: Lumpectomy, axillary block dissection, breast conserving surgery; Other: Radiotherapy

INTERVENTIONS:
Procedure: Lumpectomy, axillary block dissection, breast conserving surgery — Wide excision of primary tumor (using 1 cm surgical margins). Minimally invasive biopsy of the sentinel lymph node.
Other: Radiotherapy — Adjuvant radiotherapy carried out by institutional protocols.

SUMMARY:
The initial aesthetic and functional conditions are recorded with the help of the Breast Cancer Treatment Outcome Scale (BCTOS),an international validated questionnaire, and the Breast Cancer Conservative Treatment - cosmetic results (BCCT.core) validated computer software, allowing for comparison. Determination of the initial quality of life is measured with the European Organisation of Research and Treatment of Cancer - Quality of Life Questionnaire number C30-BR23 (EORTC QoL C30-BR23).

Patients then undergo surgical treatment according to institutional protocols. Following conventional marking of the orientation of the specimen, it is measured by an analytical scale.

Histological examination of the specimen will record the largest diameters, and parameters of the lymph nodes, according to the institutional protocol.

On the 4th week following surgery, assuming that wound healing is completed, patients' data are again recorded in BCTOS, BCCT.core and EORTC QoL C30-BR23. A third set of data are gained after completion of adjuvant radiotherapy, on the 8th postoperative month. Magnetic resonance imaging is performed to assess the volume of the contralateral breast.

Tumor - breast volume ratio is calculated, and matched up with cosmetic results in each quadrant, threshold value in the quadrants, above of which it is not advisable to perform conventional breast conserving surgery due to poor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* early breast cancer
* unilateral tumor
* tumor size is less than 3 cm

Exclusion Criteria:

* age over 70
* malignant invasive tumor in the past
* pregnancy
* previous surgical treatment of the breast or axilla
* central breast tumor sizing <3 cm
* a need for mastectomy
* tumor size >3 cm measured by mammography or physical examination
* surgical excisions resulting in positive margins
* surgical or radiotherapeutic complication

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome is the determination of the critical tumor / breast volume ratio in each quadrant, above of which number breast conserving surgery could not offer adequate cosmetic and functional results. | 8 months
  Data of eligible patients are recorded by the study physicians on a locally developed questionnaire. Digital photos are taken of each patient producing a frontal and two side views. Images are processed by the BCCT.core software (Breast Cancer Conservation Treatment. cosmetic results). Magnetic resonance imaging is implemented and used to calculate breast volume with the help of Amira 5.1 software (Visage Imaging GmbH)trial version.
  Excised tumor is measured by a validated analytical scale.

SECONDARY OUTCOMES:
Assessing the clinical applicability of the Breast Cancer Treatment Outcome Scale (BCTOS). | 8 months for each patient
  Initial cosmetic and functional status is recorded by using the validated BCTOS and the BCCT.core software.
  Patients then undergo surgical procedure according to institutional protocols. On the 4th postoperative week, patients status is recorded by BCTOS, BCTOS.core, EORTC QoL C30-BR23. After adjuvant radiotherapy (according to institutional protocols), in the 8th postoperative month, cosmetic and functional status and quality of life are assessed again with the same methods, and MR images are taken.
Assessing the relationship between cosmetic+functional results and quality of life. | 8 months for each patient
  Initial cosmetic and functional status is recorded by using the validated BCTOS and the BCCT.core software.
  Initial quality of life is assessed by the validated EORTC QoL C30-BR23. Patients then undergo surgical procedure according to institutional protocols. On the 4th postoperative week, patients status is recorded by BCTOS, BCTOS.core, EORTC QoL C30-BR23. After adjuvant radiotherapy (according to institutional protocols), in the 8th postoperative month, cosmetic and functional status and quality of life are assessed again with the same methods, and MR images are taken.
Assessing the effect of surgical intervention on cosmetic+functional results and quality of life. | During 8 postoperative months
  Initial cosmetic and functional status is recorded by using the validated BCTOS and the BCCT.core software.
  Initial quality of life is assessed by the validated EORTC QoL C30-BR23. Patients then undergo surgical procedure according to institutional protocols. On the 4th postoperative week, patients status is recorded by BCTOS, BCTOS.core, EORTC QoL C30-BR23. After adjuvant radiotherapy (according to institutional protocols), in the 8th postoperative month, cosmetic and functional status and quality of life are assessed again with the same methods, and MR images are taken.
Assessing the effect of radiotherapeutical intervention on cosmetic+functional results and quality of life. | During 8 postoperative months
  Initial cosmetic and functional status is recorded by using the validated BCTOS and the BCCT.core software.
  Initial quality of life is assessed by the validated EORTC QoL C30-BR23. Patients then undergo surgical procedure according to institutional protocols. On the 4th postoperative week, patients status is recorded by BCTOS, BCTOS.core, EORTC QoL C30-BR23. After adjuvant radiotherapy (according to institutional protocols), in the 8th postoperative month, cosmetic and functional status and quality of life are assessed again with the same methods, and MR images are taken.
Assessing the clinical applicability of the European Organisation of Research and Treatment of Cancer, Quality of Life Questionnaire C30-BR23 (EORTC QoL C30-BR23) validated questionnaire. | 8 months
  Initial quality of life is assessed by the validated EORTC QoL C30-BR23. Patients then undergo surgical procedure according to institutional protocols. On the 4th postoperative week, patients status is recorded by BCTOS, BCTOS.core, EORTC QoL C30-BR23. After adjuvant radiotherapy (according to institutional protocols), in the 8th postoperative month, cosmetic and functional status and quality of life are assessed again with the same methods, and MR images are taken.
Assessing the clinical applicability of the BCCT.core software. | 8 months
  Initial cosmetic and functional status is recorded by using the validated BCTOS and the BCCT.core software.
  Patients then undergo surgical procedure according to institutional protocols. On the 4th postoperative week, patients status is recorded by BCTOS, BCTOS.core, EORTC QoL C30-BR23. After adjuvant radiotherapy (according to institutional protocols), in the 8th postoperative month, cosmetic and functional status and quality of life are assessed again with the same methods, and MR images are taken.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Oncology, Budapest, Hungary